CLINICAL TRIAL: NCT01010048
Title: the Therapeutic Effect Treated With Tamsulosin After ESWL in Urinary Calculus
Brief Title: Compare the Therapeutic Effect Treated With Tamsulosin and Progesterone After ESWL( Extra Corporeal Shock Wave Lithotripsy) in Urinary Calculus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: He Yunfeng, The First Affiliated Hospital ,Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CQMU
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Urinary Calculus
Keywords: ESWL; urinary calculus; drugs treat
MeSH Terms: conditions — Urinary Calculi | interventions — Progesterone; Nifedipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- progesterone,tamsulosin,propantheline Bromide and nifedipine (Experimental): different effect of these drugs use to treat urinary calculus after ESWL
  Interventions: Drug: progesterone,tamsulosin,propantheline Bromide and nifedipine

INTERVENTIONS:
Drug: progesterone,tamsulosin,propantheline Bromide and nifedipine — clearance rate of stone

SUMMARY:
The purpose of this study is to compare the stone clearance rate treated with different drugs after ESWL in urinary calculus,These drugs are often used in urinary calculus,such as progesterone,tamsulosin,propantheline Bromide and nifedipine.In these study the investigators want to investigate different effect of these drugs use to treat urinary calculus after ESWL.

DETAILED DESCRIPTION:
There is 4 groups in these investigation, group1 urinary calculus treated with ESWL only ,group2 urinary calculus treated with ESWL and tamsulosin,group3 urinary calculus treated with ESWL and progesterone,group4 urinary calculus treated with ESWL ,propantheline Bromide and nifedipine.We want to investigate which one is better or not in urinary calculus treated with ESWL .

ELIGIBILITY:
Inclusion Criteria:

* From 18 years old to 68 years old,
* urinary calculus could be treated by ESWL,
* the calculus size is from 4-25mm

Exclusion Criteria:

* Less than 18 years old or more than 68 years old,
* the calculus size is from Less than4 or larger than 25mm

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
different effect of these drugs use to treat urinary calculus after ESWL | 2weeks

CONTACTS AND LOCATIONS:
Overall Officials: xiaohou wu, doctor, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital, ChongQing medical University, Chongqing, Chongqing Municipality, China